CLINICAL TRIAL: NCT05715983
Title: Comparison of Laser Destruction of Pilonidal Sinus Disease (SILAC) and Bascom
Brief Title: Comparison of Laser Destruction of Pilonidal Sinus Disease (SILAC) and Bascom II Procedure.
Acronym: SI-BAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Principal Investigator, Darya Shlyk, Russian Society of Colorectal Surgeons, Russian Society of Colorectal Surgeons
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-22
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Pilonidal Disease
Keywords: Bascom II, SiLaC, Sinus Laser Closer

STUDY DESIGN:
Intervention Model Description: assignment prospective, multi-centre.parallel-arm randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bascom II procedure (Active Comparator): Pilonidal sinus is excised, subcutaneous fat and skin are closed in the lateralization with interrupted suture.
  Interventions: Procedure: Bascom II procedure
- Sinus Laser Closer (SiLaC) (Active Comparator): Pilonidal sinus is locally excised by dermopunch or scalpel, curettage of the sinus tract with laser destruction
  Interventions: Procedure: SiLaC

INTERVENTIONS:
Procedure: Bascom II procedure — Buttocks are strapped apart with wide adhesive tape. The area is prepared using antiseptic solution twice. Solution of brilliant green with 3% hydrogen peroxide was injected in all orifices to visualize all tracts and sinuses. The proposal area of incision is marked nearby sinus tract openings and the skin with lateralization on one side of the cleft. A vertical-orientated incision of the skin and subcutaneous fat around the primary and secondary orifices is made using a scalpel or a monopolar electrocautery. The sinus tract is excised in en-block till unchanged subcutaneous tissue. The wound is irrigated with antiseptic solution. If postoperative wound is larger than 5 cm then a silicone draining tube is placed through the contraperature in the upper corner. The wound is closed by interrupted sutures Vicryl/Polysorb 2/0 3/0 layer by layer. Aseptic dressing is applied to the closed wound.
  Arms: Bascom II procedure
Procedure: SiLaC — Buttocks are strapped apart with wide adhesive tape. The area is prepared using antiseptic solution twice. Solution of brilliant green with 3% hydrogen peroxide is injected in all orifices to visualize all tracts and sinuses. All visible orifices are excised with a scalpel or dermo punch. After that hairs are removed from the sinus by Volkmann curette. A metallic stylet is used to determine the length and direction of the different tracts. Then laser destruction of the sinus is performed with FiberLase VT laser, wavelength 1460 or 1520 nm, the laser energy 10-12 Watts. The fiber delivers energy homogeneously in a continuous way. Hemostasis by electrocautery. The wound is washed with povidone-iodine solution. Aseptic dressing is applied.
  Arms: Sinus Laser Closer (SiLaC)

SUMMARY:
Surgical treatment witn lateralization of intergluteal cleft is still gold standard for pilonidal sinus disaease. But nowadays minimally invasive treatment methods such as the use of a diode laser (SiLac, Sinus Laser Closure) to obliterate the coccygeal tract are used more often. The aim of the study is to compare a new minimal invasive method (laser treatment) with traditional method ( Bascom II) in terms of recurrence rate, complications and patients satisfaction with results.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD): is 26 cases per 100,000 population, affects primarily young adults. One of the problems of surgical treatment of PSD is the frequent development of recurrence. There are various methods of surgical treatment, but the recurrence rate still high up to 67%.

Nowadays, minimally invasive methods for PSD (e.g. the use of a diode laser for sinus obliteration- SiLac, Sinus Laser Closure) compete with traditional methods. This "day-surgery" method significantly reduces the risk of postoperative complications, allows a quicker return to normal daily activity, preserves the intergluteal cleft and provides the best cosmetic results. According to some authors, the recurrence rate in this method is up to 26%, parallel others- recurrence rate is less 3 %, but the follow-up does not exceed 2 years.

On the other hand, the excision of the PSD with the mobilization of the skin-subcutaneous flap, which leads to the lateralization of the postoperative scar to one side of the intergluteal cleft hereby providing a low recurrence rate (up to 4%) .

Thus, despite the increased use of minimally invasive surgery, excision of the pilonidal sinus disease cannot be undoubtedly abandoned due to the lack of comparative studies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Chronic primary or recurrent pilonidal sinus at the remission stage.
3. Presence or absence of secondary orifices.
4. Planned surgical treatment with excision of pilonidal sinus.
5. Location of the orifices should not be less than 1 cm.
6. Location of secondary orifices less 2 cm from the natal cleft.
7. Distance between bilateral symmetrical positions of secondary orifices should not be more than 2 cm.
8. Length of the sinus in the greatest dimension, according to the ultrasound of the soft tissue of the sacrococcygeal region, should not exceed 7 cm.
9. Sinus diameter (width) in the greatest dimension should not exceed 3 cm, according to the ultrasound of the soft tissues of the sacrococcygeal region.
10. Sinus must be located directly under the skin, according to the ultrasound findings.
11. Lack of fixation of the cavity to the coccyx, when evaluating data on pelvic contrast-enhanced magnetic resonance imaging (MRI)

    ____ Non-inclusion criteria

1. Acute pilonidal sinus abscess 2. The secondary openings (orifice) position more than 3 cm from the midline. 3. Length of the cavity in the greatest dimension, according to the results of ultrasound examination, exceeds 6 cm 4. Width (diameter) of the sinus in the greatest dimension, according to the results of the ultrasound, more than 3 cm.

5. ASA > III. 6. Predictable impossibility of following the protocol 7. Pregnancy

_____ Exclusion criteria

1. The patients lost for the follow-up 2. The patient's refusal to continue participate in the investigation. 3. Impossibility of the operation performing in the planned scope

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Reccurance rate | starting from 6 months after surgery and up to 3 years after surgery]
  clinical picture of pilonidal sinus and/or appearance of new openings in the intergluteal cleft and/or chronic unhealing wound and/or residual cavity in the wound area as confirmed by the soft tissue ultrasound)

SECONDARY OUTCOMES:
Operative time | 1 day
  The length of surgery in minutes
Bloodloss | 1 day
  The amount of blood lost during surgery
Postoperative pain intensity | On 1st, 3rd, 5th and 7th postoperative day]
  early postoperative period Pain intensity will be evaluated twice a day (in the morning and in the evening) with a patient-reported Visual Analog Scale (VAS) that ranges from 0 to 10 with 0 representing no pain and 10 representing intolerable pain. A total score will be recorded.
Postoperative pain intensity - late postoperative period | On 10th, 14th, 21st, 30 day after surgery]
  Pain intensity will be evaluated once a day with a patient-reported Visual Analog Scale (VAS) that ranges from 0 to 10 with 0 representing no pain and 10 representing intolerable pain. A total score will be recorded.
Surgical site infection rate | Frame: 3 month after surgery
  The rate of infectious inflammation of the wound as confirmed by the observing doctor
Overall quality of life | 1- 7 days after surgery, 1 month, 3 months, 1 year, 3 years, 5 years after surgery
  Assessed with patient-reported questionnaire SF-12. A total score in each of 8 sections will be calculated and transformed into a 0-100 scale with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disability
Secondary surgery rate | 3 years after surgery
  The rate of surgical procedures after initial surgery performed for recurrent disease and/or wound complications
Wound healing speed | 3 years after surgery
  The time period between surgery and complete healing of the wound
Wound hemorrhage rate | Within 30 days from surgery]
  The rate of hemorrhage from wound edges
Wound seroma rate | 90 days after surgery
  The rate of seroma detection in the wound area as confirmed by soft tissues ultrasound
Patient satisfaction with cosmetic results | 6 months, 1 year, 3 years
  Patient-reported with a scale 0-10, where 0 corresponds to "completely unsatisfactory" and 10 corresponds to "completely satisfactory". A total score is registered.
Inhospital stay | 30 days]
  The duration of treatment after surgery until discharge from the hospital (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Inna Tulina, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University, Moscow, Russia, 119435; Petr Tsarkov, Prof., Study Director — I.M. Sechenov First Moscow State Medical University Moscow, Russia, 119435
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No